CLINICAL TRIAL: NCT00072839
Title: A Pilot Study of the Safety and Efficacy of ALX-0600 in Subjects With Moderately Active Crohn's Disease
Brief Title: Safety and Efficacy of ALX-0600 in Subjects With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL0600-008
Record Dates: First submitted 2003-11-11; First posted 2003-11-13 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — ALX-0600; teduglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): placebo solution injected subcutaneously daily into either thigh or abdomen.
  Interventions: Drug: placebo
- teduglutide 0.05 (Experimental): teduglutide 0.05 mg/kg/d injected subcutaneously daily.
  Interventions: Drug: Teduglutide 0.05 dose
- teduglutide 0.1 (Experimental): 0.1 mg/kg/d teduglutide injected subcutaneously into thigh or abdomen
  Interventions: Drug: teduglutide 0.1 mg dose
- teduglutide (Experimental): 0.2 mg/kg/d teduglutide injected subcutaneously into thigh or abdomen
  Interventions: Drug: ALX-0600; Drug: teduglutide 0.05; Drug: teduglutide 0.2 mg

INTERVENTIONS:
Drug: ALX-0600 — teduglutide
  Other Names: GATTEX
  Arms: teduglutide
Drug: placebo — placebo solution injected subcutaneously
  Arms: Placebo
Drug: teduglutide 0.05 — 0.05 mg/jg/d subcutaneous daily injection into thigh or abdomen
  Other Names: GATTEX
  Arms: teduglutide
Drug: teduglutide 0.2 mg — 0.2 mg/kg/d subcutaneously injected into thigh or abdomen
  Other Names: GATTEX
  Arms: teduglutide
Drug: Teduglutide 0.05 dose — 0.05 mg/kg/d subcutaneous daily injection into thigh or abdomen
  Other Names: GATTEX
  Arms: teduglutide 0.05
Drug: teduglutide 0.1 mg dose — 0.1 mg/kg/d daily subcutaneous injection into thigh or abdomen
  Other Names: GATTEX
  Arms: teduglutide 0.1

SUMMARY:
The purpose of the study is to determine whether an investigational compound, ALX-0600, is safe and effective in treating Crohn's Disease.

DETAILED DESCRIPTION:
The study is twelve weeks in duration and there are eight weeks of once-daily injections into your abdomen or thigh. There are a total of six visits.

ELIGIBILITY:
Inclusion Criteria

1. Men and women, 18 years of age and older
2. Signed and dated informed consent to participate before any study-related procedures are performed
3. Diagnosis of Crohn's disease for at least 6 months that has been documented and confirmed
4. A Crohn's Disease Activity Index (CDAI) score of 220 to 450 inclusive
5. Female subjects who are not surgically sterile or postmenopausal must use medically acceptable methods of birth control during and for 30 days after the treatment period.
6. HCT 30% or greater
7. WBC 3.5 x 109/L or greater
8. Platelets 100 x 109/L or greater
9. Adequate renal function defined as: serum creatinine and BUN 1.5 x ULN or less
10. Adequate hepatic function defined as: ALT/SPGT, AST/SGOT 2.0 x ULN or less; total bilirubin 1.25 x ULN or less, alkaline phosphatase 1.5 x ULN or less
11. Female subjects of childbearing potential must have negative urine pregnancy test results prior to randomization
12. A stool sample must be taken at screening and analyzed by a local laboratory for enteric pathogens, pathogenic ova and parasites, and Clostridium difficile toxin, and reported negative prior to randomization.
13. C-reactive protein value must be 1.0 mg/dL or more, unless there are obvious manifestations of currently active Crohn's disease such as positive observations on endoscopy, other positive indications by laboratory test results, or the subject has had a previous intestinal resection for Crohn's disease.

Exclusion Criteria

1. Nutritionally compromised subjects requiring enteral or parenteral therapy to maintain weight
2. Body weight less than 40 kg or more than 100 kg
3. Bowel obstruction or any condition that may predispose to its development, intestinal perforation, or significant gastrointestinal hemorrhage
4. Current ileostomy or colostomy or extensive external fistulization (more than 3 external fistulae which are expressible with gentle compression)
5. Expected to require surgical therapy for Crohn's disease or Crohn's disease related complications within 12 weeks of screening. If an abscess is present, it should be drained at least 3 weeks before pre-screening
6. History of ulcerative colitis within 6 months of screening visit
7. Cushing's syndrome
8. Known HIV infection, or symptoms or signs of HIV infection
9. Acute systemic infection and/or intestinal infection requiring antibiotic therapy at time of screening or baseline
10. Evidence of chronic hepatitis B or C viral infection
11. Decompensated liver disease
12. Clinically significant ECG abnormalities
13. History of angina or cardiac arrhythmia requiring drug or device intervention or clinically significant congestive heart failure or other clinically significant cardiac disease
14. History of myocardial infarction within 12 months of screening
15. History of thromboembolic disease (e.g., phlebitis, pulmonary embolus) or known congenitally or acquired prothrombotic disorder (e.g., protein C deficiency)
16. History of cancer (other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer) or clinically significant lymphoproliferative disease with fewer than 5 years documented disease-free state
17. Known substance abuse in the previous 2 years
18. Nursing mothers or pregnant women
19. Use of native GLP-2, growth hormone, or growth factors within 3 months of signing informed consent
20. Use of any of the prior or concomitant medications described in section 5.4, except as specified
21. Known hypersensitivity to any of the active or inactive constituents of ALX-0600

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-11-12 (Actual); Primary Completion 2005-07-28 (Actual); Study Completion 2005-07-28 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the percentage of subjects who respond to treatment, defined as the percentage of subjects who are in remission (CDAI less than 150) or have a 100-point or greater reduction from baseline in CDAI score at dosing Week 8. | 8 weeks of treatment

SECONDARY OUTCOMES:
The various secondary efficacy variables are based on the CDAI, Inflammatory Bowel Disease Questionnaire (IBDQ), plasma citrulline and laboratory inflammatory markers. | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (26):
- United States (21):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Rx Trials, Washington D.C., District of Columbia
  - Clinical Trials Management of Boca Raton, Boca Raton, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Venture Research, North Miami Beach, Florida
  - Visions Clinical Research - Sarasota, Sarasota, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Pinnacle Trials, Atlanta, Georgia
  - Saint Joseph's Health System, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asher Kornbluth, MD, PC, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny General Hospital-Allegheny Ctr for Digestive Diseases, Pittsburgh, Pennsylvania
  - Methodist Hospital/Baylor University, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - McGuire DVAMC, Richmond, Virginia
  - Dean Foundation Research Center, Madison, Wisconsin
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Odyssey Research, Victoria, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences, Halifax, Nova Scotia
  - Life Screening Centres, Toronto, Ontario

REFERENCES:
- [Background] Buchman AL, Katz S, Fang JC, Bernstein CN, Abou-Assi SG; Teduglutide Study Group. Teduglutide, a novel mucosally active analog of glucagon-like peptide-2 (GLP-2) for the treatment of moderate to severe Crohn's disease. Inflamm Bowel Dis. 2010 Jun;16(6):962-73. doi: 10.1002/ibd.21117. PMID 19821509